CLINICAL TRIAL: NCT06826924
Title: A Study of 7-days Water-only Fasting in Patients With Metastatic Prostate Cancer
Brief Title: 7-Days Water-Only Fasting Trial in Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Abott Lingo Wearables (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2487; IRB00456089 (Other: JHM IRB)
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Prostate Cancer
Keywords: fasting
MeSH Terms: conditions — Prostatic Neoplasms; Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fasting (Experimental): 7-day water-only fast followed by a 3-day refeeding
  Interventions: Behavioral: Fasting

INTERVENTIONS:
Behavioral: Fasting — 7 days of water-only fasting

SUMMARY:
Activating the immune system to kill cancer cells is a promising therapeutic strategy for some patients with cancer. Unfortunately, current immune-targeting treatments do not work for patients with prostate cancer. In animal models of cancer, fasting can reprogram the body's metabolism and immune cell function to help immune cells kill cancer cells. The purpose of this study is to determine whether 7 days of water-only fasting or a very low-calorie diet is safe and feasible for patients with metastatic prostate cancer. This will help the investigators develop future studies to test whether incorporating periods of fasting or very low calorie diets into treatment plans for prostate cancer can improve outcomes from this disease.

DETAILED DESCRIPTION:
Seven days of water-only fasting is safe and feasible in healthy adults. Fasting enhances anti-tumor immunity in animal models of cancer. The primary objective of this study is to determine if 7 days of water-only fasting or a ketogenic very low-calorie diet is safe and feasible in patients with metastatic prostate cancer. Patients with metastatic prostate cancer will be instructed to perform a 7-day water-only fast followed by a 3-day refeeding protocol to evaluate safety and feasibility. Eligible patients are those with metastatic prostate adenocarcinoma. Patients will perform a 7-day water-only fast followed by a 3-day refeeding protocol. Patients will be monitored by regular labs and a clinic visit on Day 3. Patients may deviate to a ketogenic very low-calorie diet at any time between Day 1 and Day 7.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
2. Age ≥18 years
3. Diagnosis of metastatic adenocarcinoma of the prostate
4. Must have a soft tissue metastasis amenable to biopsy
5. Prostate-specific antigen (PSA) is not currently declining, as determined by most recent 2 measurements taken at least 1 week apart in previous 2 months.
6. BMI between 20 and 35 kg/m2
7. Prior treatment with any prostate cancer therapy is permitted if >2 weeks from last dose. Patients are not required to have received prior treatment for prostate cancer.
8. Prior treatment with steroids is permitted if >2 weeks from last dose. Patients who cannot be weaned off steroids are not eligible.
9. Acceptable liver function:

   1. Bilirubin < 2.5 times institutional upper limit of normal (ULN)
   2. Aspartate transaminase (AST) (SGOT) and Alanine transaminase (ALT) (SGPT) < 2.5 times ULN
10. Acceptable renal function: glomerular filtration rate (GFR) of 50 mL/min/1.73 m2 or higher. GFR will be estimated by the 2021 chronic kidney disease epidemiology (CKD-EPI) creatinine equation1 using the online calculator found on UpToDate.com
11. Acceptable hematologic status:

    1. Absolute neutrophil count (ANC) ≥ 1500 cells/mm3 (1.5 ×109/L)
    2. Platelet count ≥ 100,000 platelet/mm3 (100 ×109/L)
    3. Hemoglobin ≥ 8 g/dL.
12. Acceptable electrolyte and acid/base status:

    1. Sodium 135-148 millimoles (mM) per litre
    2. Potassium 3.5-5.1mM
    3. Carbon Dioxide 21-31mM
    4. Phosphorus 2.7-4.5mM
    5. Magnesium ≥1.6mM
    6. Lactate ≤2mM
13. Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

1. ECOG Performance status ≥2
2. Unintentional weight loss greater than or equal to 5% in previous 3 months
3. Diabetes mellitus, defined as HbA1c ≥6.5% or use of medications for diabetes
4. Active uncontrolled infection. Patients with a history of HIV/AIDS may be eligible if cluster of differentiation 4 (CD4)+ T cell counts are ≥ 350 cell/ul, the patient have had no opportunistic infection within the past 12 months, the patient have been on established antiretroviral therapy (ART) for at least four weeks, and the HIV viral load is less than 400 copies/ml prior to enrollment. Patients with a history of hepatitis C virus (HCV) infection are eligible if the patient have completed curative antiviral treatment and the HCV viral load is below the limit of quantification.
5. Use of immunosuppressive medications including steroids
6. Use of diuretics or beta blockers
7. History of cardiac arrythmia, myocardial infarction, valvular heart disease, or pulmonary hypertension
8. Abnormal screening EKG
9. Daily alcohol consumption
10. Any condition or mental impairment that may compromise the ability to give informed consent, patient's safety or compliance with study requirements as determined by the investigator

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-06-03 (Estimated); Study Completion 2026-06-03 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events and serious adverse events (SAEs) | 1 year
  Number of adverse events and serious adverse events (SAEs) assessed according to CTCAE v5.0
Number patients who complete 7 days of fasting or the ketogenic very low-calorie diet of all enrolled patients | 1 year
  Number patients who complete 7 days of fasting or the ketogenic very low-calorie diet of all enrolled patients

SECONDARY OUTCOMES:
Changes in quality of life and function using Functional Assessment of Cancer Therapy - General (FACT-G) survey | Screening and daily from Day 1 to Day 10
  Changes in quality of life and function during the study based on the change in score of a daily modified FACT-G survey. Score range 0-108 with a higher score indicating better quality of life and function.
Changes in quality of life and function based on number of steps | Daily from Day 1 to Day 10
  Changes in quality of life and function during the study based on the number of steps per day by an activity tracker.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Sena, MD, PhD, Principal Investigator — SKCCC Johns Hopkins Medical Institution
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States